CLINICAL TRIAL: NCT03433768
Title: Androgen Receptor (AR) mRNA Expression is Positively Associated With Live Birth in Women Undergoing In-vitro Fertilization Independently of the Type of Ovarian Response
Brief Title: Androgen Receptor mRNA Expression is Positively Associated With Live Birth in Women Undergoing IVF Independently of the Type of Ovarian Response
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, E.M. Kolibianakis, Associate Professor, Aristotle University Of Thessaloniki
Other Study IDs: UHR 13
Record Dates: First submitted 2018-01-31; First posted 2018-02-15 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Androgen Receptor Gene Overexpression; Normal Responders; Poor Ovarian Response; Bologna Criteria
MeSH Terms: interventions — Real-Time Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- poor responders
  Interventions: Genetic: Real time PCR
- normal responders
  Interventions: Genetic: Real time PCR

INTERVENTIONS:
Genetic: Real time PCR — We take peripheral blood sample at day one, six and ten of ovarian stimulation and measure mRNA expression of androgen receptor.

SUMMARY:
AR is a steroid hormone receptor that regulates various genes' expression and affects cellular proliferation and differentiation. Androgens interact with AR, exert their paracrine action on granulosa cells and regulate gonadotropin synthesis, follicle development, oocyte maturation and corpus luteum function. Estrogens increase AR mRNA and testosterone binding site in uterine endometrium and leiomyoma. In human cancer cells, low estradiol increases AR levels, suggesting the estrogen/androgen ratio as a predictor of sex steroid response. AR mRNA expression is, also, regulated by progesterone. Although AR mRNA is expressed in the female reproductive tissues, its expression has never been studied in peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

* Women with poor ovarian response according to bologna criteria

  1. Advanced maternal age (≥40 years) or any other risk factor for poor ovarian response
  2. A previous poor ovarian response (≤3 oocytes with a conventional stimulation protocol)
  3. Abnormal ovarian reserve test, (AFC ˂5-7 follicles or AMH ˂0.5-1.1 ng/ml).
* Women with normal ovarian response with normal menstrual cycles, normal astral follicle count and normal hormonal assay.

Exclusion Criteria:

* Not more than 43 years old.
* No history of malignancies, endometriosis or polycystic ovary syndrome.
* Underlying genetic cause of infertility
* History of severe cardiac, hepatic or renal disease.
* History of systemic disease or treatment during the last three (3) months
* Participation in another interventional study and a likelihood of being unavailable for follow-up.

Ages: 20 Years to 42 Years | Sex: Female
Age Groups: Adult
Study Population: Forty normal responders and twenty-seven poor responders according to Bologna criteria, undergoing IVF/ICSI. Ovarian stimulation was performed with 200 IU recombinant follicle stimulating hormone (rFSH) and gonadotrophin releasing hormone (GnRH) antagonists. Triggering of final oocyte maturation was performed by recombinant human chorionic gonadotrophic (rhCG)
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2014-09-14 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Androgen Receptor mRNA expression | day one, six and ten of ovarian stimulation
  The expression of androgen receptor mRNA in peripheral blood of normal and poor responders level of expression in peripheral blood according to the Delta-Delta-Ct (ddCt) Algorithm.
  Percentage of increase?

SECONDARY OUTCOMES:
Serum LH levels in peripheral blood of normal and poor responders | day one, six and ten of ovarian stimulation
  level of hormone in international unit.
Serum progesterone levels in peripheral blood of normal and poor responders. | day one, six and ten of ovarian stimulation
  level of hormone in international unit.
Serum estradiol levels in peripheral blood of normal and poor responders | day one, six and ten of ovarian stimulation
  level of hormone in international unit.

IPD SHARING:
Plan to Share IPD: Undecided